CLINICAL TRIAL: NCT06420869
Title: Investigation of the Effect of Thoracic Kyphosis on Posture, Proprioception and Perception of Postural Appearance in Young Individuals
Brief Title: Investigation of the Effect of Thoracic Kyphosis Proprioception
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, sena ozdemir, Assist. Prof., Istanbul Medipol University Hospital
Other Study IDs: MedipolFTROPZ
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-05

CONDITIONS: Kyphosis; Proprioception; Posture
MeSH Terms: conditions — Kyphosis | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: The study group 1, comprised 23 subjects, comprising both males and females, with an age range of between 18 and 25 years. The subjects exhibited a thoracic kyphosis angle of ≥40° and had not undergone treatment for kyphosis in the previous six months.
  Interventions: Diagnostic Test: Assessment
- Group 2: The study group 2, comprised 23 subjects, comprising both males and females, with an age range of between 18 and 25 years.The subjects were selected based on the criteria that their thoracic kyphosis angle was less than 40° and that they did not exhibit any spinal deformities.
  Interventions: Diagnostic Test: Assessment

INTERVENTIONS:
Diagnostic Test: Assessment — A postural evaluation will be conducted, including the measurement of the thoracic kyphosis angle and the assessment of sagittal head posture.A proprioception evaluation will be conducted, whereby the cervical region, trunk and ankle joint position sense and trunk and foot sensation will be evaluated for the purpose of assessing the proprioception of the spine.Turkish adaptation of the Kyphosis Specific Spine Appearance Questionnaire (KSAQ) will be employed to assess postural appearance perception. The KSAQ is a reliable and valid patient-reported outcome tool for assessing individual perception of various aspects of kyphotic deformity and appearance in young patients with kyphosis. KSAQ is a 10-item questionnaire based on a five-point Likert scale, with responses ranging from 1 to 5. The mean of the responses is used to obtain a total score for the KSAQ. The questionnaire is related to patients' perception of appearance, with higher scores indicating a worsening of the deformity.

SUMMARY:
Although the negative effect of increased thoracic kyphosis in elderly individuals has been reported in the literature, the effect of the thoracic kyphosis angle on trunk and foot proprioception in young individuals has not been investigated. The aim of this study was to investigate the effect of the thoracic kyphosis on posture, proprioception and perception of postural appearance in young individuals.

DETAILED DESCRIPTION:
The term kyphosis is defined as an increase in the anterior curvature of the spine in the sagittal plane. Along with cosmetic deformity, individuals may experience pain with movement, increased forward head posture, unequal shoulder levels and fatigue. Kyphosis occurs when people with insufficient general muscle strength are in an upright position and high external stress is applied to the spine. Kyphosis is frequently seen in young people and children due to the demands of their school programmes and prolonged and non-ergonomic sitting positions. The prevalence of thoracic kyphosis has been reported to be 15.3% in children aged 11 years, 35% in individuals aged 20-64 years, and 38% in individuals aged 20-50 years.

The ability to perceive body positions in space without visual inputs is determined by the proprioceptive sense. Proprioceptive data from muscles, ligaments and joints contribute to the awareness of the relative orientation of the functional units of the spine at rest and in motion, enabling the control of posture and balance. Since proprioception is fundamental for movement, posture and balance, joint position sensory information from the trunk is essential for the production of synchronised muscle contractions during spinal movements. Therefore, a decrease in proprioception information may lead to an increase in the degree of kyphosis. In the literature, a negative relationship between joint position sense and the angle of kyphosis of the thoracic region has been reported in elderly individuals with thoracic kyphosis. It has been suggested that alignment problems of the spine may be related to the lack of position sense.

Over time, young people may become accustomed to inappropriate postures and poor postural awareness. Changes in posture can lead to differences in the sense of touch. These differences consist of posture-related changes in the structural properties of the skin. When dorsal skin tension increases with spinal flexion, the tactile sensitivity threshold, the longitudinal spatial acuity threshold and the transversal stretch sensitivity threshold increase. In addition, the dorsal skin decreased the sensitivity threshold to longitudinal stretch stimuli, again due to spinal flexion-induced skin tension. This suggests that sensitivity to skin stretching in a direction parallel to the spine increases as individuals move from a normal position to flexion. Changes in the flexion and extension positions of the spine produce large changes in skin stiffness, tension and thickness.

Changes in posture affect the load distribution of the foot function. A shift in the body axis away from the midline causes asymmetric loading of the extremities and affects the disproportion of the postural muscles, thus shifting the centre of gravity. Changes in the position of the trunk with deviations in the centre of gravity cause changes in the plantar load distribution with the hip and ankle. Pressure in the plantar region stimulates receptors in that region. Sensory feedback from the plantar region is important for perceiving changes in postural position and controlling postural oscillations. Feedback from cutaneous mechanoreceptors contributes functionally to proprioception of postural position and support status. However, there is a relationship between the magnitude of the kyphosis angle and the distribution of lower extremity ground reaction forces. In this context, the distribution of plantar pressure affects the sensory sensitivity of the sole of the foot.

In the forward head posture, the flexion moment of the spine is increased by maintaining the weight of the head in front of the gravity line. There is a functional and mechanical correlation between kyphosis and a forward-head posture. This position of the head can lead to further postural deviations in the body, such as rounded shoulders and increased thoracic kyphosis, in order to compensate for the deviated gravity line. This leads to a vicious circle of further deformity. The angle of the shoulder and the craniovertebral angle are negatively correlated with the forward head position and positively correlated with the sagittal head angle.

Although the negative effect of increased thoracic kyphosis in elderly individuals has been reported in the literature, the effect of the thoracic kyphosis angle on trunk and foot proprioception in young individuals has not been investigated. The aim of this study was to investigate the effect of the thoracic kyphosis on posture, proprioception and perception of postural appearance in young individuals.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 25 years of age
* Not being treated for kyphosis in the last 6 months

Exclusion Criteria:

* Those diagnosed with scoliosis and/or structural spinal deformity
* Those with any neurological deficit
* Those with concomitant disorders such as Scheuermann's disease, genetic diseases such as Beckwith-Wiedemann Syndrome or metabolic diseases that may affect body axis disorders
* Those with lower limb deformities
* Those with a history of spinal fracture and/or surgery and/or shoulder joint injury
* Those with mental disorders and intellectual disabilities.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The age range of the participants was between 18 and 25 years old.
Study Population: The study will include healthy individuals aged 18 to 25 years. A power analysis was conducted to determine the number of individuals to be included in the study. A sample size of 46 individuals was determined, with 23 individuals per group. The power of the test was calculated using the G*Power 3.1 program. A similar study in the relevant literature by Fatemeh et al. (2022) calculated the effect size to be 0.991. In order to exceed the 95% value in determining the power of the study, 46 people must be included, including 23 people in groups with a significance level of 5% and an effect size of 0.991 (df=44; t=1.711). All participants will be provided with and required to sign an informed consent form, which will be based on the principle of voluntariness.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Proprioception evaluation; Evaluation of Trunk Joint Position Sensation | 10 minute
  The BASELINE brand digital goniometer (Baseline 10044E Digital Absolute + Axis Goniometer 10044E SKU: CM10044E) can be employed for the measurement of joint position sense. Prior to commencing the measurement, participants are instructed to assume four different positions in a comfortable standing position. The participants are required to perform 30° flexion, 15° extension, 15° right and left lateral flexion for an active proprioceptive positioning test with their eyes closed. Following each position, the participants are instructed to wait for three seconds and to feel the position. They then return to the upright position and are asked to return to the position they felt and measured in that position. The deviation degrees of the participants are recorded. This process is repeated three times, with the resulting degrees of deviation averaged. During the measurement, it is essential to ensure that flexion in the knees is avoided.

SECONDARY OUTCOMES:
The Body Sensation Assessment | 10 minute
  The Body Sensation Assessment is a procedure designed to evaluate the physical sensations experienced by the subject. The assessor will then proceed to touch the T4, T5 and T6 spinous processes with a monofilament. The Semmes-Weinstein monofilament kit will be employed for the purpose of sensory evaluation. The monofilament is applied at an angle of 90°C until the tip of the monofilament is curled. The areas to be tested are maintained in contact with the monofilament for a period of 1.5 seconds, after which the monofilament is removed from the skin. Subsequently, the participant is queried as to whether they perceive the sensation and is requested to provide feedback as to whether they do or do not feel it. In the monofilament kit, starting from 2.83 and continuing up to 6.65, the initial filament, 2.83, was tested. If the participant did not perceive it, the next higher level, the thicker filament, was then evaluated.
The evaluation of foot sensation | 10 min
  The sole of the foot is tested at four sites: the heel, medial arch, lateral arch and first metatarsal. The heel position was determined to be the centre of the heel at 15% of the sole length. The medial arch position is located at 15% of the arch width from the medial border. The lateral arch is defined as the projection of the medial arch. The first metatarsal position is marked at 15% of the metatarsal width from the lateral and medial borders, respectively.
  For the dorsum of the foot, a region was delineated with the proximal boundary at 15% of the length from the lateral malleoli to the fibular head and the distal boundary at 75% of the length from the lateral malleoli to the fifth metatarsal. The dorsum test sites included a proximal, middle and distal region, each marked at a distance of 10%, 50% and 90% from the proximal border of the reference region, respectively. The Semmes-Weinstein monofilament kit will be employed for the purpose of sensory evaluation.
Ankle Joint Position Sensation Evaluation | 10 min
  The baseline brand digital goniometer (Baseline 10044E Digital Absolute + Axis Goniometer 10044E SKU: CM10044E) can be utilised for the measurement of joint position sense. The participants are blindfolded in order to prevent visual notifications. For the measurement of plantarflexion and dorsiflexion, the pivot point of the digital goniometer is placed 1.5 cm below the lateral malleolus. The fixed arm is parallel to the longitudinal axis of the fibula and aligned with the fibular head, while the mobile arm is parallel to the longitudinal axis of the fifth metatarsal. Participants are asked to perform 10° dorsiflexion, 10° and 20° plantarflexion. Individuals are instructed to actively perform the desired target angles, sense the position of the ankle for three seconds, and then return to the starting position. Individuals are then asked to repeat the target angle, and the measurement is taken in this position.
Cervical Joint Position Sense Assessment | 10 min
  Cervical position sense can be evaluated by utilising a laser pointer mounted on a lightweight headband. The subject is seated in a relaxed position with their knees and hips at 90° angles, their hands placed on their knees, in front of a sheet of paper containing a coordinate plane of A2 size and 40 cm in diameter at a distance of 90 cm, positioned at eye level. The participants are requested to focus on the natural resting head position and the origin for a period of three seconds. Subsequently, the participants are instructed to perform flexion, extension, and right-left rotation movements with their eyes closed, pausing for three seconds after each position. Subsequently, the participants are instructed to attempt to return to the initial focused position as much as possible. The point at which the participant perceives the laser beam to have reached the focal starting point is marked. The procedure should be repeated three times, and the mean value should be recorded.
Postural Assessment | 5 min
  A postural assessment will be conducted using the PostureScreen Mobile application. PostureScreen Mobile represents a pioneering application for the rapid assessment of posture. It has been demonstrated to be both valid and reliable. A camera, mounted on a tripod at shoulder height, was used to photograph the subject in lateral posture while standing in a comfortable, natural position. The angles corresponding to the photograph were then calculated. The craniovertebral angle (CVA) is the angle between the line joining the tragus of the ear to C7 and the horizontal line at C7. The shoulder angle (SA) is defined as the angle between the line joining C7 to the acromion process and the horizontal line at the acromion process. The sagittal head angle (SHA) is the angle between the line joining the tragus of the ear to the canthus of the eye and the horizontal line at the tragus.
Postural Appearance Perception | 5 min
  The Kyphosis Specific Spine Appearance Questionnaire (KSAQ), adapted into Turkish, will be used to assess the perception of postural appearance. The KSAQ is a reliable and valid patient-reported outcome tool to assess individual perception of various aspects of kyphotic deformity and appearance in young patients with kyphosis. The KSAQ is a 10-item questionnaire based on a five-point Likert scale ranging from 1 to 5, with 1 being not true; 2, somewhat true; 3, true; 4, very true; and 5, completely true. For the Kyphosis Specific Spine Appearance Questionnaire, the mean of the responses is used to obtain a total score. It is related to patients' perception of appearance, with higher scores indicating worsening of the deformity.

CONTACTS AND LOCATIONS:
Overall Officials: SENA ÖZDEMİR GÖRGÜ, PhD,PT, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided